CLINICAL TRIAL: NCT00862303
Title: Study of Autologous Dendritic Cells (DC) Loaded With Autologous Tumor Lysate (DC-Vaccine) in Combination With Cytokine-Induced Killer Cell (CIK) in Patients With Renal Cell Cancer
Brief Title: DC Vaccine Therapy Combined With Cytokine-Induced Killer Cell in Treating Patients With Renal Cell Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Fuzhou General Hospital, Fuzhou General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fuzhough0938; fuzhough0938
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2009-03

CONDITIONS: Renal Cell Carcinoma
Keywords: autologous cytokine induced killer cells; dendritic cell; vaccine; renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IL-2/IFN-α (Placebo Comparator)
  Interventions: Drug: IL-2/IFN-α
- DC-CIK (Experimental)
  Interventions: Biological: DC-CIK

INTERVENTIONS:
Biological: DC-CIK — Patients receive autologous dendritic cells (DC) loaded with autologous tumor lysate (DC vaccine) by endermic injection and infusion of CIK cells.
  Other Names: 1
  Arms: DC-CIK
Drug: IL-2/IFN-α — Patients receive treatment of IL-2 or IFN-α.
  Other Names: 2
  Arms: IL-2/IFN-α

SUMMARY:
The purpose of this study is to show if vaccination with autologous dendritic cells pulsed with tumor lysate in combination with Cytokine-Induced Killer Cell (CIK) can induce a measurable immune response in patients with renal cell carcinoma, and to evaluate the clinical effect of the regimen.

DETAILED DESCRIPTION:
The purpose of this study is to show if vaccination with autologous dendritic cells pulsed with tumor lysate in combination with Cytokine-Induced Killer Cell (CIK) can induce a measurable immune response in patients with renal cell carcinoma, and to evaluate the clinical effect of the regime.

Primary

1. Determine the clinical responses(objective response, progression-free survival, and overall survival) in patients with renal cell carcinoma treated with autologous dendritic cells (DC) loaded with autologous tumor lysate (DC vaccine) in combination with Cytokine-Induced Killer Cell (CIK).

Secondary

1. Determine cellular immune response response in terms of immuknow assay, and correlate immune response with objective clinical response in patients treated with this regimen.
2. Determine safety of multiple administrations of this regimens in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven renal cell carcinoma
* Age: > 18
* WHO- ECOG Performance Status 0-1
* At least one measurable tumor lesions according to the RECIST criteria.
* Life expectancy more than 3 months
* Written informed consent

Exclusion Criteria:

* Patients with a history of any other neoplastic disease less than 5 years ago (excepting treated carcinomas in situ of the cervix and basal/squamous cell carcinomas of the skin).
* Patients with metastatic disease in the central nervous system (CNS).
* Patients with other significant illness including severe allergy, asthma, angina pectoris or congestive heart failure.
* Patients with acute or chronic infection including HIV.
* Patients who are pregnant or nursing.
* Patients who have received antineoplastic therapy including chemotherapy or immunotherapy less than 4 weeks before beginning the trial.
* Patients who receive corticosteroids or other immunosuppressive agents.
* Patients with active autoimmune diseases such as lupus erythematosus, rheumatoid arthritis or thyroiditis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-03; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Objective tumor response (complete and partial response), Time to recurrence (TTR), Progression-free(PFS) and overall survival(OS) as measured by RECIST criteria. | every 3 months

SECONDARY OUTCOMES:
Immunity as measured by T-cell functionality (immuknow assay )to the tumor. Safety as measured by NCI common toxicity table （CTC） at completion of study. | at screening, baseline, weeks 4 , 12 and years 1 after first vaccination, and at completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Tan, M.D., Principal Investigator — Fuzhou General Hospital
Locations (1):
- Fuzhou General Hospital, Fuzhou, Fujian, China